CLINICAL TRIAL: NCT01420640
Title: Tai Chi and Aerobic Exercise for Fibromyalgia
Brief Title: Tai Chi and Aerobic Exercise for Fibromyalgia (FMEx)
Acronym: FMEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AT006367-01A1 (NIH); 1R01AT006367-01A1 (NIH)
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Tai Chi; mind-body exercise; aerobic exercise; exercise; pain
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Active Comparator)
  Interventions: Behavioral: Lower frequency, shorter period of Tai Chi; Behavioral: Higher frequency, shorter period of Tai Chi; Behavioral: Shorter frequency, longer period of Tai Chi; Behavioral: Higher frequency, longer period of Tai Chi
- Aerobic Exercise Training (Active Comparator)
  Interventions: Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Lower frequency, shorter period of Tai Chi — 12 weeks of supervised Tai Chi classes, 1x/week
  Arms: Tai Chi
Behavioral: Higher frequency, shorter period of Tai Chi — 12 weeks of supervised Tai Chi classes, 2x/week
  Arms: Tai Chi
Behavioral: Shorter frequency, longer period of Tai Chi — 24 weeks of supervised Tai Chi classes, 1x/week
  Arms: Tai Chi
Behavioral: Higher frequency, longer period of Tai Chi — 24 weeks of supervised Tai Chi classes, 2x/week
  Arms: Tai Chi
Behavioral: Aerobic Exercise Training — 24 weeks of supervised aerobic exercise training, 2x/week
  Arms: Aerobic Exercise Training

SUMMARY:
The investigators will conduct a large randomized controlled trial comparing the effectiveness of Tai Chi mind-body exercise and standard-of-care aerobic exercise for fibromyalgia. In addition, the investigators will determine the optimal frequency and duration of a Tai Chi intervention for short and long-term effectiveness.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic musculoskeletal pain syndrome that causes substantial physical and psychological impairment and costs over $25 billion annually. Current pharmacological therapies may be expensive, cause serious adverse effects, and fail to effectively improve pain and function. Finding new and effective non-pharmacological treatments for FM patients is urgently needed.

We propose to conduct the first comparative effectiveness trial of Tai Chi vs. aerobic exercise (a recommended component of the current standard of care) and to evaluate effectiveness under different Tai Chi dosing schedules in a large FM population. We aim to (1) demonstrate that, compared to aerobic exercise, Tai Chi is a more effective intervention for managing the pain and improving the functional limitations that impact quality of life for FM patients, and 2) determine the optimal frequency and duration of a supervised Tai Chi intervention in relation to short and long-term effectiveness. To achieve this goal, we will conduct a single-blind, randomized controlled trial of Tai Chi vs. aerobic exercise in 216 patients who meet the American College of Rheumatology criteria for FM. Patients will be randomized to one of four Tai Chi intervention groups: 12 or 24 weeks of supervised Tai Chi given once or twice per week, or a supervised aerobic exercise control: 2x/week for 24 weeks. All groups will have a 52-week follow-up. The primary outcome will be the FM Impact Questionnaire total score at 24 weeks. Secondary outcomes include the measures of widespread pain, functional performance, psychological functioning, self-efficacy, sleep quality, and quality of life at 12, 24, and 52 weeks.

Successful completion of the proposed study will determine the ideal regimen of Tai Chi and demonstrate that Tai Chi can be a simple, effective, and durable treatment for this therapeutically challenging disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older.
* Fulfills the American College of Rheumatology (ACR) 1990 classification criteria for FM: (1) a history of widespread musculoskeletal pain on the right and left sides of the body as well as above and below the waist for a minimum duration of 3 months, and (2) pain in 11 or more of 18 specific tender points with moderate or greater tenderness reported upon digital palpation.27
* Fulfills the ACR 2010 diagnostic criteria for FM: (WPI ≥7 AND SS ≥5) OR (WPI 3-6 AND SS ≥9) and does not have a disorder that would otherwise explain the pain28
* Willing to complete the 12-week or 24-week study, including once or twice-a-week exercise sessions.
* Willing to abstain from Tai Chi or other new formalized exercise programs until completion of the study if randomized to the Aerobic Exercise.
* Willing to abstain from Aerobic Exercise or other new formalized exercise programs until completion of the study if randomized to Tai Chi

Exclusion Criteria:

* Prior experience with Tai Chi or other similar types of Complementary and Alternative Medicine in the past 1 year such as Qi gong and yoga since these share some of the principles of Tai Chi.
* Dementia, neurological disease, cancer, cardiovascular disease, pulmonary disease, metabolic disease, renal disease, liver disease, or other serious medical conditions limiting ability to participate in the Tai Chi or Aerobic Exercise programs, as determined by the study physicians.
* Any other diagnosed medical condition known to contribute to FM symptomatology that is not under adequate control for the study period such as thyroid disease, inflammatory arthritis, systemic lupus erythematosus, rheumatoid arthritis, myositis, vasculitis or Sjogren's syndrome.
* Inability to pass the Mini-Mental Status examination (with a score below 24) 29
* Enrollment in any other clinical trial within the last 30 days
* Plan to permanently relocate from the region during the trial period
* Positive urine pregnancy test at baseline or planning pregnancy within the study period
* Not English-Speaking: English is the only language to be used during the exercise training program. Our self-reported outcome measures are obtained from validated English-version questionnaires. In addition, using other languages would likely require separate classes, recruitment and instructors which are beyond our current study scope

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire (FIQ) from baseline to 24 weeks | Week 0, Week 24
  Overall severity of FM, intensity of pain, physical function, fatigue, morning tiredness, depression, anxiety, job difficulty, and overall well-being

SECONDARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire at follow-up | Week 0, Week 12, Week 52
  Overall severity of FM, intensity of pain, physical function, fatigue, morning tiredness, depression, anxiety, job difficulty, and overall well-being
FM Symptom Severity Scale | Week 0, Week 12, Week 24, Week 52
  FM symptoms
Body Mass Index (BMI) | Week 0, Week 12, Week 24, Week 52
  General health
Medical Outcome Study Short Form 36 (SF-36) | Week 0, Week 12, Week 24, Week 52
  General health/functional status
Patient Global Assessment | Week 0, Week 12, Week 24, Week 52
  General health/functional status
The Beck Depression Inventory II | Week 0, Week 12, Week 24, Week 52
  Depression
The Chronic Pain Self-Efficacy Scale (CPSS) | Week 0, Week 12, Week 24, Week 52
  Chronic pain
The Pittsburg Sleep Quality Index (PSQI) | Week 0, Week 12, Week 24, Week 52
  Sleep quality
The Sleep Quality Numeric Rating Scale (NRS) | Week 0, Week 12, Week 24, Week 52
  Sleep quality
6-Minute Walk | Week 0, Week 12, Week 24, Week 52
  Walking ability and Endurance
The Chair Stand Test | Week 0, Week 12, Week 24, Week 52
  Physical functioning
The brief Outcome Expectation Scale (OES) | Week 0, Week 12, Week 24, Week 52
  Outcome expectations
Health Assessment Questionnaire (HAQ) | Week 0, Week 12, Week 24, Week 52
  Healthcare cost and utilization
PROMIS Health Assessment Questionnaire (HAQ) | Week 0, Week 12, Week 24, Week 52
  Health status
Muscle Strength/Power and Balance | Week 0, Week 12, Week 24, Week 52
  Physical functioning as assessed by muscle strength and power, and balance
CHAMPS Activities Questionnaire for Older Adults | Week 0, Week 12, Week 24, Week 52
  Activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wang C, Collet JP, Lau J. The effect of Tai Chi on health outcomes in patients with chronic conditions: a systematic review. Arch Intern Med. 2004 Mar 8;164(5):493-501. doi: 10.1001/archinte.164.5.493. PMID 15006825
- [Background] Wang C, Roubenoff R, Lau J, Kalish R, Schmid CH, Tighiouart H, Rones R, Hibberd PL. Effect of Tai Chi in adults with rheumatoid arthritis. Rheumatology (Oxford). 2005 May;44(5):685-7. doi: 10.1093/rheumatology/keh572. Epub 2005 Mar 1. No abstract available. PMID 15741197
- [Background] Wang C, Schmid CH, Hibberd PL, Kalish R, Roubenoff R, Rones R, McAlindon T. Tai Chi is effective in treating knee osteoarthritis: a randomized controlled trial. Arthritis Rheum. 2009 Nov 15;61(11):1545-53. doi: 10.1002/art.24832. PMID 19877092
- [Background] Wang C, Schmid CH, Rones R, Kalish R, Yinh J, Goldenberg DL, Lee Y, McAlindon T. A randomized trial of tai chi for fibromyalgia. N Engl J Med. 2010 Aug 19;363(8):743-54. doi: 10.1056/NEJMoa0912611. PMID 20818876
- [Derived] Park M, Bannuru RR, Price LL, Harvey WF, Driban JB, Wang C. Effective recruitment strategies in an exercise trial for patients with fibromyalgia. Trials. 2021 Aug 21;22(1):557. doi: 10.1186/s13063-021-05502-3. PMID 34419131
- [Derived] Wang C, Schmid CH, Fielding RA, Harvey WF, Reid KF, Price LL, Driban JB, Kalish R, Rones R, McAlindon T. Effect of tai chi versus aerobic exercise for fibromyalgia: comparative effectiveness randomized controlled trial. BMJ. 2018 Mar 21;360:k851. doi: 10.1136/bmj.k851. PMID 29563100
- [Derived] Wang C, McAlindon T, Fielding RA, Harvey WF, Driban JB, Price LL, Kalish R, Schmid A, Scott TM, Schmid CH. A novel comparative effectiveness study of Tai Chi versus aerobic exercise for fibromyalgia: study protocol for a randomized controlled trial. Trials. 2015 Jan 30;16:34. doi: 10.1186/s13063-015-0548-x. PMID 25633475